CLINICAL TRIAL: NCT00450242
Title: Use of 5% Lidocaine Ointment in the Treatment of Vulvar Vestibulitis
Brief Title: 5% Lidocaine Ointment in the Treatment of Vulvar Vestibulitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05-2332
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-06

CONDITIONS: Vulvar Vestibulitis
Keywords: vulvar vestibulitis; vestibulitis
MeSH Terms: conditions — Vulvar Vestibulitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% Lidocaine cream (Experimental): 5% topical lidocaine cream.
  Interventions: Drug: 5% topical lidocaine ointment
- Placebo cream (Placebo Comparator)
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: 5% topical lidocaine ointment — Lidocaine 5% in hydrophilic petrolatum, dime-sized amount, applied nightly.
  Arms: 5% Lidocaine cream
Drug: Placebo cream — hydrophilic petrolatum, dime-sized amount, applied nightly.
  Arms: Placebo cream

SUMMARY:
* Study Hypothesis: Use of 5% topical lidocaine ointment will result in improved ability to have sexual intercourse and decreased pain scores in women with vestibulitis when compared to placebo.
* This is a study to assess if topical lidocaine will improve symptoms in women with vulvar vestibulitis. It compares use of nightly 5% topical lidocaine ointment to placebo ointment. The duration of the study is 8 weeks. 28 women will be in each arm for a total of 56 women in the study.

DETAILED DESCRIPTION:
* After consent is obtained patients will undergo the following treatment plan: randomization to treatment with 5% lidocaine ointment or placebo for vestibulitis. There will be 56 women total (28 in each arm).The placebo used will be hydrophilic petrolatum. Randomization will be performed using computer generated permuted blocks. A standard history and physical exam incorporating assessment of skin allodynia (testing with q-tip swab) on the vestibule and pressure measurements of the pelvic floor muscles (how much tenderness there is on perineal muscles with palpation) will be performed. Baseline questionnaires that will evaluate sexual frequency, sexual function survey (Female sexual function index), the modified Gracely pain scale of intercourse related pain, and psychometric evaluation including evaluation of anxiety, somatization (State-Trait Anxiety Inventory and Brief Symptom Inventory). Depression can also be evaluated with the Brief Symptom Inventory. Lastly, overall quality of health can be assessed with the SF-12. There is a baseline, 2 week and 6 week visit. Women will abstain from intercourse during these 6 weeks. Women will have a physical exam evaluation of the vestibule at each visit. They will then be able to have intercourse and will repeat surveys of sexual frequency, function, pain scale of intercourse related pain and the SF-12 at 8 weeks.
* Aim 1: To assess if lidocaine ointment produces a superior treatment response to placebo.
* Hypothesis 1: Use of topical lidocaine, compared with placebo, will result in improved sexual function and self-reported pain scores. This is to be measured as the ability to have successful intercourse. Secondarily, sexual function, quality of life and scores for intercourse related pain will be evaluated.
* Aim 2: To assess if there are predictors of response to treatment such as demographics, duration of disease, primary or secondary vulvar vestibulitis, or psychometric assessments (anxiety and somatization).
* Hypothesis 2: There are predictors of response to treatment of vulvar vestibulitis based upon patient characteristics, characteristics of the disease and psychometric assessments.

ELIGIBILITY:
Inclusion Criteria:

* women with the clinical diagnosis of vvs who have dyspareunia as their primary complaint. They must have a current sexual partner.

Exclusion Criteria:

* postmenopausal
* pure vaginismus
* generalized vulvodynia
* pudendal neuralgia
* pregnant, breastfeeding
* less than 2 months post delivery
* diagnosis of dermatologic condition on biopsy
* positive fungal culture
* currently on treatment for vvs
* history of lidocaine treatment for vvs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Rohl, MD, Study Director — UNC Division of Advanced Laparoscopy and Pelvic Pain; Denniz Zolnoun, MD MPH, Principal Investigator — UNC- Division of Advanced Laparoscopy and Pelvic Pain; John Steege, MD, Study Chair — UNC Division of Advanced Laparoscopy and Pelvic Pain
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 subjects were recruited via advertisement and clinical referrals from within the medical center and from the community of referring physicians.
Period: Overall Study
Arm/Group | 5% Lidocaine Cream | Placebo Cream
Started | 7 | 7
Completed | 4 | 6
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Lidocaine Cream | Placebo Cream | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.9 (8.5) | 29.4 (5.7) | 29.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Report the Ability to Have Intercourse
Description: Participants' response upon inquiry.
Time Frame: baseline, week 8
Population: Three lidocaine subjects and one control subject failed to complete the study.
Measure: Number; unit: participants
Groups:
- Placebo Cream: Topical cream vehicle.
Arm/Group | 5% Lidocaine Cream | Placebo Cream
Number analyzed (Participants) | 4 | 6
participants | 4 | 6

2. Primary Outcome: Change in Visual Analog Scale (VAS) Scores With Intercourse From Baseline to Week 8
Description: Visual Analog Scale (VAS) scores (range 0-100 mm; 0 = none, 100 = worst pain) were recorded for pain during intercourse during baseline and week 8 of the study, for lidocaine treated subjects and controls. The "mean" listed for each group is average week 8 score subtracted from the average baseline score.
Time Frame: baseline, week 8
Population: three lidocaine subjects and one control subject failed to complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5% Lidocaine Cream | Placebo Cream
Number analyzed (Participants) | 4 | 6
units on a scale | 2.5 (10.3) | 19.7 (24.3)

3. Secondary Outcome: SF-12 Quality of Life Scores
Description: The SF-12 is a subset of 12 items from the Medical Outcomes Study 36-Item Short Form Survey (SF-36) and was collected at the bi-weekly office visits. Each score ranges from 0-100. The components measure physical and mental health, respectively. Higher scores are indicative of better function. ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, and age.
Time Frame: baseline, week 8
Population: The study terminated due to lack of funding and difficulties with recruitment. More extensive data analysis to include secondary outcome measures was not performed due to inability to fund statistical programming and analysis efforts.
Measure: Number; unit: units on a scale
Arm/Group | 5% Lidocaine Cream | Placebo Cream
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Modified Gracely Pain Scale
Description: The Modified Gracely Pain Scale consists of two components: 1) three numerical scales scored 0-100 for lowest, average, and highest pain level during during the preceding week, and 2) two word choice scales measuring affective and intensity levels. Each word in the word choice scales has an assigned number. Change scores on each subscale can thus be calculated over time (baseline v. week 8).
Time Frame: baseline, week 8
Population: as for outcome 3
Measure: Number; unit: units on a scale
Arm/Group | 5% Lidocaine Cream | Placebo Cream
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 5% Lidocaine Cream | Placebo Cream
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6

LIMITATIONS AND CAVEATS:
The study terminated due to lack of funding and difficulties with recruitment. More extensive data analysis to include secondary outcome measures was not performed due to inability to fund statistical programming and analysis efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes